CLINICAL TRIAL: NCT03148769
Title: Spanish Cohort of Bacteriemias 2016: Epidemiology, Clinical Management and Prognostic Factors at Diagnosis.
Brief Title: Spanish Bacteriemia Cohort 2016: Epidemiology, Clinical Management and Prognosis Factors
Acronym: PRO-BAC
Status: Completed | Type: Observational
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Collaborators: Hospital Universitario Virgen Macarena (Other)
Responsible Party: Sponsor
Other Study IDs: FIS-AMO-2016-01
Record Dates: First submitted 2017-04-05; First posted 2017-05-11 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Bacteremia
Keywords: Bloodstream infections, epidemiology
MeSH Terms: conditions — Bacteremia; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Microbial strains
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Bacteremia

The Hypothesis of the study are the followings:

* To demonstrate relevant epidemiologic and clinical changes with potentially impact in the management and prognosis of the patients with bacteremia.
* Since the diagnosis and management is heterogeneous between centers, we could identify a scenario to improve.
* To identify quality indicators in the management of bacteremia.
* To demonstrate that some interventions made by Bacteremia Team pose relevant impact in the prognosis of bacteremia.

ELIGIBILITY:
Inclusion Criteria:

* Every episode of bacteremia in patients older than 13 years old, confirmed microbiologically and clinically significant (presence of clinical sepsis data at diagnosis) should be prospectively included on the basis of standard criteria.
* Episodes of transient bacteremia may be included.
* Drugs will be prescribed in the usual way, according to the conditions established in the authorization. The assignment of a patient to a particular therapeutic strategy will not be decided in advance by the study protocol, but will be determined by the usual clinical practice, and the decision to prescribe a particular drug will be clearly dissociated from the decision to include to the patient in the study.

Exclusion Criteria:

* Bacteremias without clinical relevance

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: It will be included all episodes of bacteremia diagnosed over a year in all participating hospitals in patients over 13 years old. It´s no possible to make a calculation of the sample size, this will depend on the type of hospital, the number of beds of the same and the number of blood cultures that are requested during the period of recruitment of the study.
Sampling Method: Non-Probability Sample
Enrollment: 5320 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Epidemiology and prognostic factors of bacteremia episodes. | From day 0 to day 30
  * Global incidence and per type of acquisition.
  * Global etiology and per type of acquisition.
  * Frequency of multiresistant and emerging microorganism.
  * Source of bacteremia.
  * Clinical severity of presentation.
  * Clinical failure, mortality at day 7, mortality at day 30, recurrence, length of stay and re-admission at hospital.

SECONDARY OUTCOMES:
Clinical management of patients with bacteremia during the episode. | From day 0 to day 30
  * Antibiotic therapy used during the episodes (empirical and targeted).
  * Non antibiotic therapy/support therapy used during the episode.
  * Frequency of focus search and adequate control.
Differences in the management between types of services, wards and hospitals. | From day 0 to day 30
  Comparison between different services and hospital wards of variables regarding on the management of episodes.
Influence of clinical management in the prognosis. | From day 0 to day 30
  - Identifying prognostic factors related with mortality, clinical failure and recurrence.
Developing and validating a predictive model for early and late mortality. | From day 0 to day 30
  - Developing and validating a predictive model for mortality based in prognostic factors related with mortality.
Quality indicators in the management of bacteremia. | From day 0 to day 30
  - Identifying quality indicators in the management of episodes of bacteremia.
Interventions made by Bacteremia Team. | From day 0 to day 30
  * Frequency and type of interventions made by Bacteremia Teams.
  * Impact of these interventions in the management and prognosis of episodes.

CONTACTS AND LOCATIONS:
Overall Officials: Jesús Rodríguez-Baño, MD PhD, Study Director — Unidad Clínica de Enfermedades Infecciosas, Microbiología. Hospital Universitario Virgen Macarena
Locations (29):
- Spain (29):
  - Public Health Agency Business Hospital de Poniente., El Ejido, Almería
  - General Hospital of Granollers, Granollers, Barcelona
  - University Hospital Mútua de Terrasa, Terrassa, Barcelona
  - Hospital Punta Europa, Algeciras, Cádiz
  - Jerez de la Frontera Hospital, Jerez de la Frontera, Cádiz
  - Hospital San Juan de la Cruz, Úbeda, Jaen
  - Hospital El Bierzo, Ponferrada, León
  - Costa del Sol Hospital, Márbella, Málaga
  - University Hospital of Vigo, Vigo, Pontevedra
  - University General Hospital of Alicante, Alicante
  - Torrecárdenas Hospital, Almería
  - L´ Esperit Sant ( Santa Coloma Granemet) Hospital, Barcelona
  - University Hospital of Burgos, Burgos
  - University Hospital Puerta del Mar, Cadiz
  - La Linea de la Concepción Hospital, Cadiz
  - Puerto Real Hospital, Cadiz
  - University Hospital Reina Sofía, Córdoba
  - University Hospital San Cecilio, Granada
  - University Hospital Virgen de las Nieves, Granada
  - Ciudad de Jaén Hospital, Jaén
  - University Hospital of León, León
  - University Hospital Arnau de Vilanova, Lleida
  - University Hospital Carlos Haya ( Málaga), Málaga
  - Central University Hospital of Asturias, Oviedo
  - University Clinic of Navarra, Pamplona
  - University Hospital Marqués de Valdecilla, Santander
  - University Hospital Virgen Macarena, Seville
  - University Virgen de Valme Hospital, Seville
  - Universitary Hospital Cruces, Vizcaya

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Garnacho-Montero J, Garcia-Garmendia JL, Barrero-Almodovar A, Jimenez-Jimenez FJ, Perez-Paredes C, Ortiz-Leyba C. Impact of adequate empirical antibiotic therapy on the outcome of patients admitted to the intensive care unit with sepsis. Crit Care Med. 2003 Dec;31(12):2742-51. doi: 10.1097/01.CCM.0000098031.24329.10. PMID 14668610
- [Result] Vincent JL, Sakr Y, Sprung CL, Ranieri VM, Reinhart K, Gerlach H, Moreno R, Carlet J, Le Gall JR, Payen D; Sepsis Occurrence in Acutely Ill Patients Investigators. Sepsis in European intensive care units: results of the SOAP study. Crit Care Med. 2006 Feb;34(2):344-53. doi: 10.1097/01.ccm.0000194725.48928.3a. PMID 16424713
- [Result] Rodriguez-Bano J, Lopez-Prieto MD, Portillo MM, Retamar P, Natera C, Nuno E, Herrero M, del Arco A, Munoz A, Tellez F, Torres-Tortosa M, Martin-Aspas A, Arroyo A, Ruiz A, Moya R, Corzo JE, Leon L, Perez-Lopez JA; SAEI/SAMPAC Bacteraemia Group. Epidemiology and clinical features of community-acquired, healthcare-associated and nosocomial bloodstream infections in tertiary-care and community hospitals. Clin Microbiol Infect. 2010 Sep;16(9):1408-13. doi: 10.1111/j.1469-0691.2009.03089.x. PMID 19845694
- [Result] Lopez-Cortes LE, Del Toro MD, Galvez-Acebal J, Bereciartua-Bastarrica E, Farinas MC, Sanz-Franco M, Natera C, Corzo JE, Lomas JM, Pasquau J, Del Arco A, Martinez MP, Romero A, Muniain MA, de Cueto M, Pascual A, Rodriguez-Bano J; REIPI/SAB group. Impact of an evidence-based bundle intervention in the quality-of-care management and outcome of Staphylococcus aureus bacteremia. Clin Infect Dis. 2013 Nov;57(9):1225-33. doi: 10.1093/cid/cit499. Epub 2013 Aug 8. PMID 23929889
- [Result] Pappas PG, Kauffman CA, Andes D, Benjamin DK Jr, Calandra TF, Edwards JE Jr, Filler SG, Fisher JF, Kullberg BJ, Ostrosky-Zeichner L, Reboli AC, Rex JH, Walsh TJ, Sobel JD; Infectious Diseases Society of America. Clinical practice guidelines for the management of candidiasis: 2009 update by the Infectious Diseases Society of America. Clin Infect Dis. 2009 Mar 1;48(5):503-35. doi: 10.1086/596757. PMID 19191635
- [Result] Rodriguez-Bano J, Pano-Pardo JR, Alvarez-Rocha L, Asensio A, Calbo E, Cercenado E, Cisneros JM, Cobo J, Delgado O, Garnacho-Montero J, Grau S, Horcajada JP, Hornero A, Murillas-Angoiti J, Oliver A, Padilla B, Pasquau J, Pujol M, Ruiz-Garbajosa P, San Juan R, Sierra R; Grupo de Estudio de la Infeccion Hospitalaria-Sociedad Espanola de Enfermedades Infecciosas y Microbiologia Clinica; Sociedad Espanola de Farmacia Hospitalaria; Sociedad Espanola de Medicina Preventiva, Salud Publica e Higiene. [Programs for optimizing the use of antibiotics (PROA) in Spanish hospitals: GEIH-SEIMC, SEFH and SEMPSPH consensus document]. Enferm Infecc Microbiol Clin. 2012 Jan;30(1):22.e1-22.e23. doi: 10.1016/j.eimc.2011.09.018. Epub 2011 Dec 15. Spanish. PMID 22178010
- [Result] Mosier MJ, Ton-That H. Making the case for de-escalation therapy in ventilator-associated pneumonia once again. Crit Care Med. 2013 Jul;41(7):1810-1. doi: 10.1097/CCM.0b013e31828ce949. No abstract available. PMID 23774344
- [Result] Kaye KS. Antimicrobial de-escalation strategies in hospitalized patients with pneumonia, intra-abdominal infections, and bacteremia. J Hosp Med. 2012;7 Suppl 1:S13-21. doi: 10.1002/jhm.983. PMID 23737333
- [Result] Gaynes R. Health care--associated bloodstream infections: a change in thinking. Ann Intern Med. 2002 Nov 19;137(10):850-1. doi: 10.7326/0003-4819-137-10-200211190-00015. No abstract available. PMID 12435223
- [Result] Cisneros-Herreros JM, Sanchez-Gonzalez M, Prados-Blanco MT, Llanos-Rodriguez C, Vigil-Martin E, Soto-Espinosa de los Monteros B, Pachon-Diaza J. [Blood cultures in the emergency department]. Enferm Infecc Microbiol Clin. 2005 Mar;23(3):135-9. doi: 10.1157/13072162. Spanish. PMID 15757584
- [Result] Fridkin SK, Hageman JC, Morrison M, Sanza LT, Como-Sabetti K, Jernigan JA, Harriman K, Harrison LH, Lynfield R, Farley MM; Active Bacterial Core Surveillance Program of the Emerging Infections Program Network. Methicillin-resistant Staphylococcus aureus disease in three communities. N Engl J Med. 2005 Apr 7;352(14):1436-44. doi: 10.1056/NEJMoa043252. PMID 15814879
- [Result] Rodriguez-Bano J, Navarro MD, Romero L, Martinez-Martinez L, Muniain MA, Perea EJ, Perez-Cano R, Pascual A. Epidemiology and clinical features of infections caused by extended-spectrum beta-lactamase-producing Escherichia coli in nonhospitalized patients. J Clin Microbiol. 2004 Mar;42(3):1089-94. doi: 10.1128/JCM.42.3.1089-1094.2004. PMID 15004058
- [Result] Al-Hasan MN, Juhn YJ, Bang DW, Yang HJ, Baddour LM. External validation of bloodstream infection mortality risk score in a population-based cohort. Clin Microbiol Infect. 2014 Sep;20(9):886-91. doi: 10.1111/1469-0691.12607. Epub 2014 Mar 26. PMID 25455590
- [Result] Al-Hasan MN, Lahr BD, Eckel-Passow JE, Baddour LM. Predictive scoring model of mortality in Gram-negative bloodstream infection. Clin Microbiol Infect. 2013 Oct;19(10):948-54. doi: 10.1111/1469-0691.12085. Epub 2012 Nov 27. PMID 23190091
- [Result] Retamar P, Portillo MM, Lopez-Prieto MD, Rodriguez-Lopez F, de Cueto M, Garcia MV, Gomez MJ, Del Arco A, Munoz A, Sanchez-Porto A, Torres-Tortosa M, Martin-Aspas A, Arroyo A, Garcia-Figueras C, Acosta F, Corzo JE, Leon-Ruiz L, Escobar-Lara T, Rodriguez-Bano J; SAEI/SAMPAC Bacteremia Group. Impact of inadequate empirical therapy on the mortality of patients with bloodstream infections: a propensity score-based analysis. Antimicrob Agents Chemother. 2012 Jan;56(1):472-8. doi: 10.1128/AAC.00462-11. Epub 2011 Oct 17. PMID 22005999
- [Result] Retamar P, Lopez-Prieto MD, Natera C, de Cueto M, Nuno E, Herrero M, Fernandez-Sanchez F, Munoz A, Tellez F, Becerril B, Garcia-Tapia A, Carazo I, Moya R, Corzo JE, Leon L, Munoz L, Rodriguez-Bano J; Sociedad Andaluza de Enfermedades Infecciosas/Sociedad Andaluza de Microbiologia y Parasitologia Clinica and Red Espanola de Investigacion en Enfermedades Infecciosas (SAEI/SAMPAC/REIPI) Bacteremia Group; Rodriguez-Lopez F, Garcia MV, Fernandez-Galan V, del Arco A, Perez-Santos MJ, Sanchez Porto A, Torres-Tortosa M, Martin-Aspas A, Arroyo A, Garcia-Figueras C, Acosta F, Florez C, Navas P, Escobar-Lara T. Reappraisal of the outcome of healthcare-associated and community-acquired bacteramia: a prospective cohort study. BMC Infect Dis. 2013 Jul 24;13:344. doi: 10.1186/1471-2334-13-344. PMID 23883281
- [Result] Retamar P, Lopez-Prieto MD, Rodriguez-Lopez F, de Cueto M, Garcia MV, Gonzalez-Galan V, Del Arco A, Perez-Santos MJ, Tellez-Perez F, Becerril-Carral B, Martin-Aspas A, Arroyo A, Perez-Cortes S, Acosta F, Florez C, Leon-Ruiz L, Munoz-Medina L, Rodriguez-Bano J; SAEI/SAMPAC/REIPI Bacteremia Group. Predictors of early mortality in very elderly patients with bacteremia: a prospective multicenter cohort. Int J Infect Dis. 2014 Sep;26:83-7. doi: 10.1016/j.ijid.2014.04.029. Epub 2014 Jul 5. PMID 25008770
- See also: European Surveillance of Antimicrobial Consumption Network (ESAC-Net). — http://ecdc.europa.eu/en/publications/Publications/antimicrobial-consumption-europe-esac-net-2012.pdf